CLINICAL TRIAL: NCT07117721
Title: Evaluation of Endoscopic Band Ligation for Treatment of Type 2 Diabetes: A Single-Center Interventional Study
Brief Title: Endoscopic Band Ligation for Type 2 Diabetes Mellitus (ENDOBAND-DM)
Acronym: ENDOBAND-DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: El Katib Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abeid, Consultant Gastroenterologist and Bariatric Endoscopist, Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M.Abeid-ENDOBAND-DM-2025
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Endoscopic band ligation; Duodenal intervention; Metabolic endoscopy; GLP-1; GIP; Insulin resistance; HbA1c; Non-surgical diabetes treatment; Duodenal mucosal modulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Single-center prospective pilot study. All enrolled participants will undergo endoscopic band ligation in the second through fourth parts of the duodenum and be followed for metabolic outcomes over 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENDOBAND-DM (Experimental): Participants in this arm will undergo endoscopic band ligation (ENDOBAND-DM) targeting the second through fourth parts of the duodenum, from just distal to the ampulla of Vater to the ligament of Treitz. The procedure is designed to induce localized mucosal changes that may enhance enteroendocrine signaling (e.g., GLP-1, GIP) and improve glycemic control in patients with type 2 diabetes mellitus.
  Interventions: Procedure: Endoscopic Band Ligation (ENDOBAND-DM)

INTERVENTIONS:
Procedure: Endoscopic Band Ligation (ENDOBAND-DM) — Endoscopic band ligation of the second through fourth parts of the duodenum, from just distal to the ampulla of Vater to the ligament of Treitz. The aim is to induce localized mucosal remodeling that may enhance enteroendocrine signaling (GLP-1, GIP) and improve glycemic control in patients with type 2 diabetes mellitus.
  Other Names: ENDOBAND - DM; Duodenal Banding

SUMMARY:
This is a pilot clinical study evaluating the safety and feasibility of Endoscopic Band Ligation (ENDOBAND-DM) applied to the second through fourth parts of the duodenum - from just distal to the ampulla of Vater to the ligament of Treitz - in patients with type 2 diabetes mellitus (T2DM). The goal is to induce mucosal remodeling in this duodenal segment, potentially enhancing gut hormone signaling and improving glycemic control. Participants will be monitored for changes in HbA1c, fasting glucose, and insulin sensitivity over 6-12 months.

DETAILED DESCRIPTION:
The duodenum is a key site of nutrient sensing and hormonal regulation, and duodenal dysfunction contributes to the pathophysiology of type 2 diabetes mellitus (T2DM).

This single-center prospective pilot study investigates Endoscopic Band Ligation (ENDOBAND-DM) targeting the second through fourth parts of the duodenum, beginning just distal to the ampulla of Vater and extending to the ligament of Treitz.

The endoscopic application of elastic bands is designed to induce localized mucosal changes in the duodenum, potentially modulating enteroendocrine responses such as GLP-1 and GIP secretion and improving insulin sensitivity.

Adult participants with suboptimally controlled T2DM (HbA1c 7.5-10.5%) who are not on insulin therapy will undergo a single EBL session. Follow-up will occur at 1, 3, 6, and 12 months post-intervention.

Primary outcome: Change in HbA1c at 6 months. Secondary outcomes include changes in fasting glucose, insulin resistance indices (e.g., HOMA-IR), gut hormones, weight, and adverse events.

This study introduces a novel endoscopic approach aimed at duodenal mucosal modulation for metabolic benefit in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Confirmed diagnosis of type 2 diabetes mellitus
* HbA1c between 7.5% and 10.5% at screening
* Body Mass Index (BMI) between 27 and 40 kg/m²
* Stable use of oral antidiabetic medications for ≥3 months prior to enrollment
* Willingness to undergo endoscopic procedure and attend all follow-up visits
* Signed informed consen

Exclusion Criteria:

* Use of insulin therapy
* Previous bariatric or gastrointestinal surgery
* Diagnosis of type 1 diabetes mellitus
* Known gastrointestinal obstruction, ulcers, or active GI bleeding
* History of pancreatitis, biliary disease, or abnormal anatomy in duodenum
* Pregnancy or breastfeeding
* Severe comorbidities (e.g., uncontrolled cardiovascular disease, advanced kidney or liver disease)
* Use of GLP-1 receptor agonists within 3 months prior to enrollment
* Inability or unwillingness to comply with the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c level from baseline | Baseline and 6 months post-intervention
  Mean change in glycosylated hemoglobin (HbA1c) will be measured at 6 months after the endoscopic band ligation procedure, compared to baseline values. This will assess the primary glycemic effect of the intervention.

SECONDARY OUTCOMES:
Change in fasting plasma glucose | Baseline and 6 months
  Measured in mg/dL to assess improvement in fasting glucose levels after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Abeid, MD, MSc, Principal Investigator — Faculty of Medicine, Cairo Univesity

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including baseline characteristics, intervention details, and outcome measures) will be shared with qualified researchers upon reasonable request, starting 12 months after study completion and for up to 5 years. Requests should be directed to mohamedabeid@gmail.com and will require a data access agreement.

REFERENCES:
- [Background] Yli-Hankala A. [Is my patient sleeping?]. Duodecim. 1998;114(16):1563-9. No abstract available. Finnish. PMID 11717791